CLINICAL TRIAL: NCT04439526
Title: Observational Study on GUselkumab: Effectiveness and Impact on quaLity of LIfe in naïVE or Bio Experienced Patients With Regional (Facial and Genital) Psoriasis (GULLIVER Study)
Brief Title: A Study of Guselkumab in Naive or Bio-experienced Participants With Regional (Facial and Genital) Psoriasis
Acronym: GULLIVER
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108761; CNTO1959PSO4013 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
Keywords: Facial; Genital
MeSH Terms: conditions — Psoriasis; Facies | interventions — guselkumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Facial Psoriasis: Participants with moderate facial psoriasis who are being treated with guselkumab in real world practice will be observed in this study.
  Interventions: Drug: Guselkumab
- Participants with Genital Psoriasis: Participants with moderate genital psoriasis who are being treated with guselkumab in real world practice will be observed in this study.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Participants with moderate facial and/or genital psoriasis treated with guselkumab (as prescribed by their physician) in real world practice will be observed in this study.
  Other Names: Tremfya

SUMMARY:
The purpose of this study is to investigate the effectiveness profile of guselkumab used in a real-life setting in participants with moderate facial and/or genital psoriasis. Effectiveness will be evaluated using the static Physicians Global Assessment (sPGA) for the facial region and the sPGA for the genital region.

ELIGIBILITY:
Inclusion Criteria:

Participants included in the study:

* must have a first or confirmed diagnosis of psoriasis, requiring systemic treatment with significant involvement (defined as a Static Physician's Global Assessment [sPGA] score greater than or equal to [>=] 3) involving the facial and/or genital regions
* must have started treatment according to the approved indication as described in the current version of summary of product characteristics (SmPC) of the product approved in Italy. Enrollment may occur at any time after the first injection of guselkumab but before completion of the next visit at week 4 or 12 as scheduled according to common clinical practice
* must sign an informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

Participants will be excluded from the study if they:

* have any contraindication to the use of guselkumab, as stated in the current SmPC of the product approved in Italy
* received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before the start of guselkumab treatment
* are currently enrolled in another clinical trial or investigational study
* are currently enrolled in an observational study sponsored or managed by a Janssen company
* participant unable to read, to write, to understand and sign the informed consent form (ICF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with facial and/or genital psoriasis, receiving guselkumab treatment as standard of care (SOC) in clinical practice, will be observed. The primary data source for the study will be the medical records of each participating participant.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Static Physician's Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) and at Least a 2-grade Improvement for the Facial Region | Week 52
  The sPGA for the facial region is a physician global rating of psoriasis severity, which evaluates plaque thickness, scaling and erythema, at a given point in time. The sPGA comprises a 6-point rating scale from 0 to 5 where 0 = clear, 1 = minimal/ almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
Percentage of Participants Achieving a sPGA Score of Clear (0) or Almost Clear (1) and at Least a 2-grade Improvement for the Genital Region | Week 52
  The sPGA for the genital region is a physician global ratings of psoriasis severity, which evaluates plaque thickness, scaling and erythema, at a given point in time. The sPGA comprises a 6-point rating scale from 0 to 5 where 0 = clear, 1 = minimal/ almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a sPGA Score of Clear (0) or Almost Clear (1) and at least a 2-grade Improvement for the Facial Region | Week 12, Week 28
  The sPGA for the facial region is a physician global rating of psoriasis severity, which evaluates plaque thickness, scaling and erythema, at a given point in time. The sPGA comprises a 6-point rating scale from 0 to 5 where 0 = clear, 1 = minimal/ almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
Percentage of Participants Achieving a sPGA Score of Clear (0) or Almost Clear (1) and at least a 2-grade Improvement for the Genital Region | Week 12, Week 28
  The sPGA for the genital region is a physician global rating of psoriasis severity, which evaluates plaque thickness, scaling and erythema, at a given point in time. The sPGA comprises a 6-point rating scale from 0 to 5 where 0 = clear, 1 = minimal/ almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
Change from Baseline in the Dermatology Quality of life Index (DLQI) Total Score for the Facial Region | Baseline, Week 12, Week 28, Week 52
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participants' quality of life. Each question is evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate greater impact on quality of life. The DLQI is calculated by summing the scores of the questions and ranges from 0 to 30 where 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate greater impact on quality of life of participants.
Change from Baseline in the DLQI Total Score for the Genital Region | Baseline, Week 12, Week 28, Week 52
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participants' quality of life. Each question is evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate greater impact on quality of life. The DLQI is calculated by summing the scores of the questions and ranges from 0 to 30 where 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate greater impact on quality of life of participants.
Change from Baseline in the SF-36 Physical Component Summary (PCS) Score for the Facial Region | Baseline, Week 12, Week 28, Week 52
  The SF-36 is a survey that measures 8 domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Each item is scored on a scale of 0 to 100. Worst value is 0 and best value is 100.
Change from Baseline in the SF-36 PCS Score for the Genital Region | Baseline, Week 12, Week 28, Week 52
  The SF-36 is a survey that measures 8 domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Each item is scored on a scale of 0 to 100. Worst value is 0 and best value is 100.
Change from Baseline in the SF-36 Mental Component Summary (MCS) Score for the Facial Region | Baseline, Week 12, Week 28, Week 52
  The SF-36 is a survey that measures 8 domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Each item is scored on a scale of 0 to 100. Worst value is 0 and best value is 100.
Change from Baseline in the SF-36 MCS Score for the Genital Region | Baseline, Week 12, Week 28, Week 52
  The SF-36 is a survey that measures 8 domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Each item is scored on a scale of 0 to 100. Worst value is 0 and best value is 100.
Change from Baseline in Pain/Itch/Discomfort Visual Analogue Scale (VAS) Scores for the Facial Region | Baseline, Week 12, Week 28, Week 52
  Each VAS is a patient-rated assessment designed to evaluate the intensity of pain, itch or discomfort on a linear scale of 0-100. Operationally, each VAS is represented by a 100 mm horizontal line anchored by extreme descriptors at each end, where 0 = "No Symptom" and 100 = "Worst Symptom Imaginable".
Change from Baseline in Pain/Itch/Discomfort VAS Scores for the Genital Region | Baseline, Week 12, Week 28, Week 52
  Each VAS is a patient-rated assessment designed to evaluate the intensity of pain, itch or discomfort on a linear scale of 0-100. Operationally, each VAS is represented by a 100 mm horizontal line anchored by extreme descriptors at each end, where 0 = "No Symptom" and 100 = "Worst Symptom Imaginable".
Change from Baseline in Redness/Scaling/Thickness VAS Scores for the Facial Region | Baseline, Week 12, Week 28, Week 52
  Each VAS is a patient-rated assessment designed to evaluate the intensity of redness, scaling, and thickness on a linear scale of 0-100. Operationally, each VAS is represented by a 100 mm horizontal line anchored by extreme descriptors at each end, where 0 = "No Sign" and 100 = "Worst Sign Imaginable".
Change from Baseline in Redness/Scaling/Thickness VAS Scores for the Genital Region | Baseline, Week 12, Week 28, Week 52
  Each VAS is a patient-rated assessment designed to evaluate the intensity of redness, scaling, and thickness on a linear scale of 0-100. Operationally, each VAS is represented by a 100 mm horizontal line anchored by extreme descriptors at each end, where 0 = "No Sign" and 100 = "Worst Sign Imaginable".
Percentage of Participants Achieving an Overall sPGA Score of Clear (0) or Almost Clear (1) and at least a 2-grade Improvement Among Participants with an Overall sPGA Score greater than or equal to (>=) 3 at baseline | Baseline, Week 12, Week 28, Week 52
  The overall sPGA is defined as physician global rating of psoriasis severity, which evaluates plaque thickness, scaling and erythema, at a given point in time. The sPGA comprises a 6-point rating scale from 0 to 5 where 0 = clear, 1 = minimal/ almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
Percentage of Participants Achieving a Psoriasis Area and Severity Index (PASI) 100 Response Among Participants with a PASI Score >10 at Baseline | Baseline, Week 12, Week 28, Week 52
  The PASI is a tool to assess and grade the severity of psoriasis and response to therapy. In the PASI, the body is divided into four areas: the head, trunk, upper extremities and lower extremities. Each of these areas is assessed separately for the percentage of surface area involved, which translates to a numeric score that ranges from 0 to 6, and for degree of erythema, scaling and induration/thickness, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72, with higher score indicating more severe disease status. A PASI 100 response is defined as 100 percent (%) improvement in PASI score from baseline.
Percentage of Participants Achieving a PASI 90 Response Among Participants with a PASI Score >10 at Baseline | Baseline, Week 12, Week 28, Week 52
  The PASI is a tool to assess and grade the severity of psoriasis and response to therapy. In the PASI, the body is divided into four areas: the head, trunk, upper extremities and lower extremities. Each of these areas is assessed separately for the percentage of surface area involved, which translates to a numeric score that ranges from 0 to 6, and for degree of erythema, scaling and induration/thickness, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72, with higher score indicating more severe disease status. A PASI 90 response is defined as >=90% improvement in PASI score from baseline.
Percentage of Participants Achieving a PASI 75 Response Among Participants with a PASI Score >10 at Baseline | Baseline, Week 12, Week 28, Week 52
  The PASI is a tool to assess and grade the severity of psoriasis and response to therapy. In the PASI, the body is divided into four areas: the head, trunk, upper extremities and lower extremities. Each of these areas is assessed separately for the percentage of surface area involved, which translates to a numeric score that ranges from 0 to 6, and for degree of erythema, scaling and induration/thickness, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72, with higher score indicating more severe disease status. A PASI 75 response is defined as >=75% improvement in PASI score from baseline.
Mean Percent Change in PASI Score from Baseline | Baseline, Week 12, Week 28, Week 52
  The PASI is a tool to assess and grade the severity of psoriasis and response to therapy. In the PASI, the body is divided into four areas: the head, trunk, upper extremities and lower extremities. Each of these areas is assessed separately for the percentage of surface area involved, which translates to a numeric score that ranges from 0 to 6, and for degree of erythema, scaling and induration/thickness, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72, with higher score indicating more severe disease status. Mean percent change from baseline in PASI score will be assessed.
Mean Change in Percent Body Surface Area (BSA) from Baseline in Participants with BSA >10% at Baseline | Baseline, Week 12, Week 28, Week 52
  BSA affected by psoriasis of <5% is considered mild psoriasis, 5-10% moderate psoriasis, and >10% severe psoriasis.
Percentage of Participants Achieving an Absolute PASI Score of Less Than (<) 3 Among Participants with a PASI Score of >10 at Baseline | Baseline, Week 12, Week 28, Week 52
  The PASI is a tool to assess and grade the severity of psoriasis and response to therapy. In the PASI, the body is divided into four areas: the head, trunk, upper extremities and lower extremities. Each of these areas is assessed separately for the percentage of surface area involved, which translates to a numeric score that ranges from 0 to 6, and for degree of erythema, scaling and induration/thickness, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72, with higher score indicating more severe disease status. Percentage of participants who achieve an absolute PASI score <3 will be assessed.
Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Week 52
  The TSQM-9 is a 9-item generic participant-reported outcome instrument to assess participants' satisfaction with medication and covers domains of effectiveness, convenience and global satisfaction. The instrument is scored by domain with scores ranging from 0-100, where a lower score indicates lower satisfaction.
Persistency with Guselkumab | Up to Week 52
  Persistency with treatment is defined as duration of time from initiation to last dose of therapy, as well as the percentage of participants still on treatment at the end of the observation period.
Narrative Plots at Enrollment and Week 52 | Baseline (at enrollment) and Week 52
  Participants will be invited to fill in two narrative plots; one at the enrollment visit and one at the week 52 visit.
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 52
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (38):
- Italy (38):
  - Policlinico di Bari Ospedale Giovanni XXIII, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Ospedale San Giovanni di Dio, Cagliari
  - PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania
  - Azienda Ospedaliera Universitaria - OO.RR. San Giovanni di Dio Ruggi d'Aragona, Cava de' Tirreni
  - Università D'Annunzio, Chieti
  - Azienda Ospedaliero Universitaria di Ferrara, Cona
  - Ospedale Sant'Antonio Abate, Erice
  - Azienda Sanitaria di Firenze-Ospedale Piero Palagi, Florence
  - IRCCS Aor San Martino IST, Genova
  - Ospedale San Salvatore, L’Aquila
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - AO Papardo, Messina
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Az. Ospedaliero - Universitaria di Modena, Modena
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Università del Piemonte Orientale - Ospedale Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale Maggiore, Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale S. Maria Della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Grande Ospedale Metropolitano 'Bianchi-Melacrino-Morelli' Reggio Calabria, Reggio Calabria
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - ISG San Gallicano, Roma
  - AOU Policlinico Umberto I, Roma
  - Istituto Dermopatico dell'Immacolata, Roma
  - Policinico A Gemelli, Roma
  - Policlinico Tor Vergata, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Santa Maria, Terni
  - Ospedale Alfredo Fiorini, Terracina
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
  - A.O. Universitaria Ospedali Riuniti di Ancona, Torrette Di Ancona
  - Azienda Ospedaliero Universitaria S.Maria Della Misericordia, Udine
  - Ospedale S.S. Giovanni e Paolo, Venezia

IPD SHARING:
Plan to Share IPD: No